CLINICAL TRIAL: NCT00213096
Title: A Randomized, Open-Label Study Comparing the Effect of a Contraceptive Vaginal Ring Delivering Daily Doses of 150 Micrograms Nestorone and 15 Micrograms Ethinyl Estradiol to an Oral Contraceptive Containing 150 Micrograms of Levonorgestrel and 30 Micrograms of Ethinyl Estradiol Per Tablet on Hepatic Factors Including Coagulation Factors
Brief Title: Effects of Hormonal Contraceptives on Liver Proteins and Coagulation Factors: A Comparison of a Contraceptive Vaginal Ring and an Oral Contraceptive
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Population Council #323; HRN-A-00-99-00010
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Contraception
Keywords: Contraceptive agents; female
MeSH Terms: interventions — ST 1435

INTERVENTIONS:
Drug: Nestorone/ethinyl estradiol contraceptive vaginal ring; levonorgestrel/ethinyl estradiol oral contraceptive

SUMMARY:
The purpose of this 3-month (cycle) study was to evaluate the effects of hormonal contraceptives containing a progestin and an estrogen on liver proteins and coagulation factors that are sensitive to estrogen. In this study, a contraceptive vaginal ring containing Nestorone® (a progestin with no androgenic properties) and ethinyl estradiol was compared to an oral contraceptive containing levonorgestrel (an androgenic progestin) and ethinyl estradiol.

DETAILED DESCRIPTION:
The purpose of this 3-month (cycle) study was to evaluate the effects of hormonal contraceptives containing a progestin and an estrogen on liver proteins and coagulation factors that are sensitive to estrogen. In this study, a contraceptive vaginal ring containing Nestorone® (a progestin with no androgenic properties) and ethinyl estradiol was compared to an oral contraceptive containing levonorgestrel (an androgenic progestin) and ethinyl estradiol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, aged 18-34 years, who did not wish to become pregnant for 3 months (or 5 months if first discontinuing oral contraceptives
* Intact uterus and at least 1 ovary
* Have regular menstrual cycles (28 ± 7 days) or 2 regular cycles after parturition or abortion
* Willing to use condoms while having sexual intercourse during the 3 month study (or 5 months if discontinuing oral contraceptives), or
* Willing to continue use of a specified non-hormonal method of birth control including permanent sterilization, non-hormone-containing IUD, male condoms, or abstinence during the study or to use condoms if discontinuing one of these methods
* Willing and able to comply with the protocol
* Willing and able to sign informed consent prior to entry into the study and prior to discontinuing another method of contraception
* Easy venous access

Exclusion Criteria:

* Pregnancy
* Known hypersensitivity to estrogens or progestins
* Known hypersensitivity to silicone rubber
* Undiagnosed vaginal discharge or vaginal lesions or abnormalities
* Smoking status: >15 cigarettes per day
* Breastfeeding
* Current or past thrombophlebitis or thromboembolic disorders
* Family history of venous thrombosis or embolism (1st degree relatives <55 years of age)
* Known history of Factor V Leiden or positive screening test for APC-resistance
* Current or past cerebrovascular or coronary artery disease
* Carcinoma (hormone-dependent tumor; past history of any carcinoma not in remission for >5 years)
* Medically diagnosed severe depression
* Headaches with focal neurological symptoms
* Undiagnosed abnormal genital bleeding
* History of cholestatic jaundice of pregnancy or jaundice with prior steroid use
* Benign or malignant liver tumors; active liver disease
* Diastolic/systolic BP ≥90/140 mmHg after 5 min. rest
* Known or suspected alcoholism (>2 drinks/day)or drug abuse
* Positive for hepatitis B & C and/or HIV 1 or 2, abnormal screening CBC, serum chemistry values (including fasting, total cholesterol and triglycerides), abnormal Pap smear, abnormal findings on dipstick urinalysis, or an abnormal electrocardiogram (ECG)
* Participation in a clinical trial within last 3 months or more than 1 trial in the last year
* BMI (kg/m2) >28
* Use of injectable contraceptives in last 6 months (e.g. cyclofem or DMPA)
* Unwilling to stop oral contraceptives for 2 months prior to study initiation
* Use of implanted hormonal contraceptives, including Mirena or Implanon, in last 2 years
* Not living in the catchment area of the clinic*Severe cystoceles or rectoceles

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2003-03 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Comparison of the differences between contraceptive vaginal ring and oral contraceptive treatment groups in change from baseline to end of treatment in serum angiotensinogen and sex-hormone binding globulin.

SECONDARY OUTCOMES:
Comparison of the differences between contraceptive vaginal ring & oral contraceptive treatment groups in change from baseline to end of treatment in serum or plasma concentrations of 15 other hepatic proteins, coagulation factors & coagulation markers.

CONTACTS AND LOCATIONS:
Overall Officials: Regine Sitruk-Ware, MD, Principal Investigator — Population Council
Locations (1):
- Center for Human Drug Research, Leiden, Netherlands